CLINICAL TRIAL: NCT04000139
Title: A Multi-center, Multi-national, Randomized, Double-blind, Placebo Controlled, Parallel Group, Phase IIa Study to Evaluate the Efficacy, Safety and Tolerability of an Anthocyanin-rich Extract (ACRE) in Patients With Ulcerative Colitis
Brief Title: Anthocyanin Rich Extract (ACRE) in Patients With Ulcerative Colitis
Acronym: ACRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); The Broad Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACRE
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Ulcerative Colitis
Keywords: bilberry; anthocyanin; anthocyanin-rich extract; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two treatment arms, active ingredient or placebo with the ratio 2:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized anthocyanin rich extract (Active Comparator): 3 doses of 2x 500mg in capsules daily
  Interventions: Drug: Standardized anthocyanin-rich extract
- Placebo (Placebo Comparator): 3 doses of 2x 500mg in capsules daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Standardized anthocyanin-rich extract — 3g of anthocyanin-rich extract taken daily as: 3 doses of 2x 500mg. Treatment duration 56 days (8 weeks).
  Arms: Standardized anthocyanin rich extract
Drug: Placebo — 3g of placebo taken daily as: 3 doses of 2x 500mg. Treatment duration 56 days (8 weeks).
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of a bilberry derived anthocyanin-rich extract in patients with ulcerative colitis. Two thirds of participants will receive the anthocyanin-rich extract, while one third will receive placebo, for 8 weeks of treatment.

DETAILED DESCRIPTION:
For anthocyanins (ACs), a wide range of protective biological effects have been described, such as anti-oxidative, anti-carcinogenic, anti-microbial and anti-inflammatory activities. Various research groups could identify a beneficial effect of ACs in IBD and intestinal inflammation.

A total of 112 subjects will be randomized. Subjects will be screened for eligibility between 0 and 28 days prior to baseline visit. At the baseline visit, subjects with moderate to severe ulcerative colitis (Mayo score ≥6) and fulfilling all inclusion/exclusion criteria will be randomized into two treatment arms (ACRE or placebo). Total duration of drug product administration will be 8 weeks (56 days) followed by a follow-up phase of 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Established diagnosis of UC, with minimum time from diagnosis of ≥3 months
3. Moderately at least left sided UC (disease should extend 15 cm or more above the anal verge). Disease severity determined by a Modified Mayo score of 6 to 12 with an endoscopic sub score ≥2 assessed by central reading of endoscopy performed at screening visit and no other individual sub score <1 (see 9.8.2 for more detailed information)
4. Current oral or rectal 5-ASA/SP use or a history of oral or rectal 5-ASA/SP use
5. Current steroids use or history of steroids dependency, refractory, or intolerance, including no steroids treatment due to earlier side-effects (only one of the steroids criteria have to be fulfilled, see definition in European Crohn´s and Colitis organization (ECCO) guidelines)
6. One of the following points must be fulfilled:

   1. Active disease despite induction therapy with 5-ASA agents where adequate therapy is considered with an oral 5-ASA (mesalamine 2- 4.8 g/day, sulfasalazine 4-6 g/day) administered for at least 2 weeks. Topical treatment with 5-ASA may have been attempted but this is not a prerequisite for inclusion in the study OR
   2. Intolerance to oral 5-ASAs or azathioprine OR
   3. Active disease despite a thiopurine (adequately dosed according to treatment guidelines, such as 2-3 mg/kg for azathioprine) or methotrexate administered for at least 12 weeks.
7. Allowed to receive a therapeutic dose of following UC drugs during the study:

   1. Oral steroids therapy (≤30 mg prednisone or equivalent/daily) providing that the dose has been stable for 2 weeks prior Baseline
   2. Oral or rectal MMX Budesonide therapy (9mg/daily) initiated and a stable dose at least 2 months before Baseline
   3. Oral or rectal 5-ASA/SP compounds, providing that the dose has been stable for 2 months prior to Baseline and initiated at least 8 weeks before screening.
   4. AZA/6-MP providing that the dose has been stable for 8 weeks prior to Baseline and been initiated at least 2 months before screening
   5. TNF inhibitors (Infliximab, Adalimumab or Golimumab) are allowed, providing that the dose is stable for at least 2 months prior to baseline and during the study treatment period
   6. Vedolizumab and Tofacitinib is allowed providing that the dose is stable for at least 2 months prior to baseline and during the study treatment period
8. Ability to understand the treatment, willingness to comply with all study requirements and ability to provide informed consent

Exclusion Criteria:

Subjects fulfilling any of the following criteria are not eligible for inclusion in this study:

1. Suspicion of differential diagnosis such as; Crohn's enterocolitis, ischaemic colitis, radiation colitis, indeterminate colitis, infectious colitis, diverticular disease, associated colitis, microscopic colitis, massive pseudopolyposis or non-passable stenosis
2. Acute fulminant UC and/or signs of systemic toxicity
3. UC limited to the rectum (disease which extends <15 cm above the anal verge)
4. History of malignancy, except for:

   1. Treated (cured) basal cell or squamous cell in situ carcinoma
   2. Treated (cured) cervical intraepithelial neoplasia or
   3. carcinoma in situ of the cervix with no evidence of recurrence within the previous 5 years prior to the screening visit
5. History or presence of any clinically significant disorder that, in opinion of the investigator, could impact on patient's possibility to adhere to the protocol and protocol procedures or would confound the study result or compromise patient safety
6. Long term treatment with antibiotics or non-steroidal anti-inflammatory drugs (NSAIDs) within two weeks prior to screening (one short treatment regime for antibiotics and occasional use of NSAIDS are allowed)
7. Serious active infection
8. Gastrointestinal infections including positive Clostridium difficile stool assay
9. Currently receiving parenteral nutrition or blood transfusions
10. Females who are lactating or have a positive serum pregnancy test during the screening period
11. Concurrent participation in another clinical study with investigational therapy or previous use of investigational therapy within 5 half-lives and within at least 30 days after last treatment of the experimental product prior to enrolment
12. Subjects who have been treated with

    a. A dose of ≥ 1 mg per kg body weight prednisone or ≥30mg/d in the last 4 weeks prior to randomization.
13. Ongoing treatment with cyclosporine or tacrolimus. Eligible subjects must have stopped cyclosporine and/or tacrolimus at least 4 weeks and antibiotics at least 1 week prior to randomization.
14. known history of alcohol abuse, chronic liver or biliary disease
15. Repeated and confirmed laboratory findings showing:

    1. total bilirubin greater than 2 x upper limit of the normal range (ULN) unless in context of Gilbert's syndrome
    2. alkaline phosphatase (AP) greater than 2 x ULN
    3. ALT (SGPT) greater than 2 x ULN
    4. serum creatinine greater than 2 X ULN
    5. total white blood cell count (WBC) outside the range of 3,000 - 15,000 /μL. Subjects with mild leukocytosis (WBC not higher than 15,000 /μL) may be eligible, especially if the elevated WBC, according to the Investigator, is attributable to corticosteroid therapy and other causes such as hematological or infectious diseases can be excluded.
    6. platelet count <100,000/μL
    7. Hemoglobin less 8 g/dL and/or other signs of severe anemia.
16. History or presence of a significant renal disease.
17. Significant illness within the two weeks prior to dosing or any active systemic infection or medical condition that may require treatment or therapeutic intervention during the study.
18. Current history of active systemic bacterial, viral or fungal infections
19. Presence or history of underlying metabolic, endocrine, hematologic, pulmonary, cardiac, blood, renal, hepatic, infectious, psychiatric or any medically unstable condition, as assessed by the primary treating physician which, in the opinion of the investigator, would place the subject at unacceptable risk for participation in the study.
20. Known allergies to bilberries or any other AC containing fruits
21. Planned diet change, any severe or new dietary restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Clinical response at week 8 | 8 weeks
  Proportion of patients with clinical response at week 8 where clinical response is defined as the reduction of total mayo score ≥ 3 points

SECONDARY OUTCOMES:
Clinical remission at week 8 | 8 weeks
  Proportion of patients with symptomatic clinical remission at week 8, where clinical remission is defined as total mayo score ≤ 2, with no individual sub-score > 1
Rectal bleeding | 8 weeks
  Proportion fo patients with absence of rectal bleeding at week 8, defined by the mayo subscore rectal bleeding of 0
Stool frequency | 8 weeks
  Proportion of patients with normal or enhanced stool frequency at Week 8, defined by the Mayo sub score stool frequency of 0 or 1 (with at least one point decrease from Baseline, Week 0)
Endoscopic remission | 8 weeks
  Proportion of patients with endoscopic remission at Week 8, defined by the Modified Mayo endoscopic sub score of 0 or 1 (excluding friability)
Histological remission | 8 weeks
  Proportion of patients with histological remission at Week 8, defined by the Geboes Index of grade 0 or 1
Symptomatic remission | 4 weeks
  Proportion of patients with symptomatic remission at Week 4, defined by the Mayo sub scores, i) rectal bleeding of 0, ii) stool frequency of 0 or 1 (with at least one point decrease from Baseline, Week 0), (patient reported outcome)
Rectal bleeding week 4 | 4 weeks
  Proportion of patients with absence of rectal bleeding at Week 4, defined by the Mayo sub score rectal bleeding of 0
Stool frequency week 4 | 4 weeks
  Proportion of patients with normal or enhanced stool frequency at Week 4, defined by the Mayo sub score stool frequency of 0 or 1 (with at least one point decrease from Baseline, Week 0)
Durable symptomatic remission | 8 weeks / 12 weeks
  Proportion of patients with durable symptomatic remission, defined by the Mayo sub scores, i) rectal bleeding of 0, ii) stool frequency of 0 or 1 (with at least one point decrease from Baseline, Week 0) [PRO2] at both Week 8 and Week 12
Clinical response | 8 weeks
  Proportion of patients with clinical response at Week 8, defined as clinical remission or a three point and ≥30 % decrease from Baseline, Week 0 in the sum of the Modified Mayo score, i) rectal bleeding, ii) stool frequency and iii) endoscopy score (excluding friability), iiii) physicians global assessment (PGA)
Fecal calprotectin | 8 weeks
  Mean change in fecal calprotectin at Week 1, 2, 4, and 8 compared to Baseline, Week 0.
Steroid dosage | 4 weeks (follow-up phase)
  Mean change in steroid dosage for patients in remission at Week 8 to Week 12
SIBDQ | 8 weeks
  Mean change in each of the short inflammatory bowel disease questionnaire (SIBDQ) sub domains at Week 8 compared to Baseline, Week 0 SIBDQ data will consist of 10 individual items, scores for the 4 dimensions (bowel function, emotional status, systemic symptoms and social function) and a total score. All data will be listed and data for the 4 dimensions and total score summarized by time post-dose for each dose. Week 8 changes from baseline for the 4 dimensions and total score will be plotted and summarized by dose to visually assess dose-related changes.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Rogler, Prof. Dr. med. Dr. phil., Study Director — Universitätsspital Zürich
Locations (6):
- Switzerland (6):
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern
  - Gastroenterologische Praxis Balsiger, Seibold & Partner, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No